CLINICAL TRIAL: NCT06471322
Title: A Multi-Disciplinary Technology-Based Care After Hospitalization for Diabetic Ketoacidosis in Patients With Type 1 Diabetes
Brief Title: A Multi-Disciplinary Technology-Based Care for Diabetic Ketoacidosis in Patients With Type 1 Diabetes
Acronym: DKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was too difficult - not enough patients were enrolled after 1 year
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 23-697
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis | interventions — Continuous Glucose Monitoring; Standard of Care

STUDY DESIGN:
Intervention Model Description: Control Arm: Historical group of patients admitted for DKA In the prior 1 year Intervention: Patients with type 1 diabetes mellitus admitted to the hospital with confirmed diabetic ketoacidosis treated with intra-venous insulin infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm - Standard of Care, retrospective (Other): Retrospective data looking at 12 patients undergoing standard of care for diabetic ketoacidosis
  Interventions: Other: Standard of Care
- Intervention Arm - Continuous Glucose Monitoring (CGM) (Active Comparator): 12 patients with confirmed diabetic ketoacidosis upon hospital admission will receive continuous glucose monitor (CGM)
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — Patients will wear a continuous glucose monitor upon discharge from the hospital for six months
  Arms: Intervention Arm - Continuous Glucose Monitoring (CGM)
Other: Standard of Care — Standard of Care - retrospective review
  Arms: Control Arm - Standard of Care, retrospective

SUMMARY:
The study team proposes that use of a novel multi-disciplinary approach with continuous glucose monitoring technology can significantly improve glycemic control and reduce readmissions among those with type 1 diabetes mellitus (T1DM) admitted for Diabetic ketoacidosis (DKA). This will also help promote a pathway for care of these patients after admission utilizing resources which are available within the Endocrinology, Diabetes and Metabolism department at the Cleveland Clinic.

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is a serious complication of type 1 diabetes mellitus (T1DM) with significant cost to the United States of $2.2 billion over the past decade. Readmissions are very common with a 20.2% readmission rate within 30 days of discharge and 86% of those admitted with DKA having a subsequent 1-3 admissions in the following year. While predictors have been identified (i.e. lower socioeconomic status, Medicaid/Medicare, younger age, female, leaving against medical advice, etc.), few interventions have been able to concretely show a reduction in the rate of readmission apart from endocrinology consultation. Very few studies have assessed the use of a multi-disciplinary approach in this context. The only study in adults with T1DM which made use of such a team (i.e. ketoacidosis case manager, educators to provide immediate post-discharge contact and follow up along with behavioral health, education and endocrinology follow up) was done in the UK and was able to show significant improvement in readmission and glycemic control over the year-long intervention, but notably had to shut down due to lack of funding. None of these interventions consistently applied technology (i.e. continuous glucose monitoring [CGM]) which is known to be able to significantly improve glycemic control within the first month of use in those with poorly controlled T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Diagnosis of Type 1 Diabetes
* Admitted to the hospital with confirmed diabetic ketoacidosis treated with intravenous insulin infusion
* No prior use of continuous glucose monitoring (CGM)
* Compatible smart phone with CGM
* Allergy to any component of the CGM

Exclusion Criteria:

* Condition which, in investigator judgement would limit their ability to participate safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Measure improvement in glycemic control | 6 months
  To compare improvement in glycemic control (HBA1c measured in % glycosylated hemoglobin) between baseline at hospitalization for DKA and 6 months later using CGM intervention versus standard of care.

SECONDARY OUTCOMES:
Assess change in number of readmissions | 6 months
  To assess change in number of readmissions between baseline and 6 months later using CGM intervention versus standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Keren, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No